CLINICAL TRIAL: NCT07334899
Title: The Effect of Game-Based Learning on Kinesiophobia Patient Management of Physiotherapy and Rehabilitation Students: A Randomized Controlled Investigation
Brief Title: The Effect of Game-Based Learning on Kinesiophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Assist Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NEU-PT2025-06
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Learning
Keywords: Physiotherapy; Education; learning style; game-based education; Attitude toward profession

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group interventional model in which participants were randomly allocated to a study group receiving game-based learning training on approaching patients with kinesiophobia alongside the standard curriculum, or to a control group receiving the standard curriculum only for 14 weeks.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to group allocation to minimize assessment bias. The assessor had no involvement in the intervention process and was unaware of whether participants belonged to the study or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Participants in the education group received a 14-week structured training program based on game-based learning focused on approaching patients with kinesiophobia, in addition to their standard physiotherapy curriculum. The training was delivered face-to-face and included interactive and scenario-based educational activities designed to improve students' knowledge, awareness, and clinical attitudes toward patients with kinesiophobia.
  Interventions: Other: Game-Based Learning Training on Approaching Patients With Kinesiophobia
- Control group (Experimental): Participants in the control group continued with the standard physiotherapy curriculum for 14 weeks and did not receive any additional training related to game-based learning or approaching patients with kinesiophobia during the study period.
  Interventions: Other: Routine Physiotherapy Education

INTERVENTIONS:
Other: Game-Based Learning Training on Approaching Patients With Kinesiophobia — The intervention consisted of a structured game-based learning training program designed to improve physiotherapy students' approach to patients with kinesiophobia. Each training session lasted approximately 60-90 minutes and was delivered face-to-face by the responsible researcher.
  The training included four main components: (1) a brief theoretical lecture (15-20 minutes) covering kinesiophobia, pain psychology, and patient management; (2) case-based learning (20-30 minutes) involving analysis of fictional clinical scenarios; (3) game-based and interactive activities (20-30 minutes) focused on the management of kinesiophobia; and (4) group work and discussion (15-20 minutes), during which students collaboratively solved problems and discussed scenarios tailored to varying levels of patients' psychological and physical status.
  Gamified quizzes were integrated into the training using an escape room format developed via the Genially platform. Students progressed through the activity by
  Arms: Education group
Other: Routine Physiotherapy Education — Participants in the control group continued their standard physiotherapy curriculum for the same study period. No additional training, game-based learning activities, case simulations, or kinesiophobia-specific educational content were provided during the intervention period.
  Arms: Control group

SUMMARY:
Aim:

The aim of this study was to evaluate the impact of innovative teaching methods applied in the "Physiotherapy and Innovation" course conducted during the 2024-2025 spring semester on physiotherapy students' learning experiences, and to describe the process of developing and exhibiting student-designed materials at the end of the course.

Method:

The study was carried out with 45 third-year students enrolled in the Department of Physiotherapy and Rehabilitation at Necmettin Erbakan University, Faculty of Health Sciences. The course was enriched with project-based learning, group brainstorming sessions, prototype development, presentations, and feedback meetings in line with innovative teaching principles. At the end of the semester, students designed prototypes of innovative tools, exercise materials, or educational aids applicable in the field of physiotherapy. The developed materials were presented at the "Innovative Physiotherapy Materials Exhibition" organized within the university.

DETAILED DESCRIPTION:
The use of games in health education dates back to the 1980s .The emergence of game development for improving the clinical application characteristics of products in health education. Game rules designed for education should include elements such as goals, problem-solving, critical thinking, winning ability, content, competition, and fun. Games are used in many health education fields such as formality, midwifery, physiotherapy, gerontology, pharmacology, and more. Although individual education is increasingly common in health education today, active learning methods may be preferred over traditional teaching methods. Therefore, game-based learning environments have led to better learning compared to traditional teaching methods. Openable milk cartons are available. In the field of health, in today's conditions where science and technology are rapidly centralized, and knowledge, skills, and attitudes are constantly updated, educational activities should be designed in a way that is appropriate for the age. Students can learn and teach while having fun by designing games as universal educational materials. In line with this need, in Physiotherapy and Rehabilitation education, different training methods are available in student training according to the physiotherapist's various patient approaches. The effect of determining the effect of play-based learning in the kinesiophobic game of these effective Physiotherapy and Rehabilitation centers is still being determined.

ELIGIBILITY:
Inclusion Criteria:

* Being a physiotherapy and rehabilitation student
* Volunteering to participate in the study
* For the education group, volunteering to participate in the game-based learning training on approaching patients with kinesiophobia

Exclusion Criteria:

* Inability to understand, read, or communicate in Turkish
* Failure to participate in any stage of the study (e.g., pre-test, in-class education session, or post-test)
* Requesting withdrawal from the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
The Attitudes Toward the Physiotherapy Profession Scale | From enrollment to the end of the 14-week training period
  The Attitudes Toward the Physiotherapy Profession Scale, developed by Turhan in 2018, is a 35-item, five-point Likert-type instrument. Thirty-three items are scored from 1 (strongly disagree) to 5 (strongly agree), while two items (items 26 and 30) are reverse scored. Total scores range from 35 to 175, with higher scores indicating more positive attitudes toward the physiotherapy profession.
  The scale consists of three subscales: professional satisfaction, required professional qualifications, and general professional concerns. The Kaiser-Meyer-Olkin measure of sampling adequacy was 0.833, and Bartlett's test of sphericity was significant (χ² = 10058.592, p < 0.001). The overall Cronbach's alpha coefficient was 0.977, with subscale alpha values of 0.966, 0.974, and 0.957, respectively. Pearson correlation coefficients were 0.96, 0.91, and 0.90 for the subscales and 0.92 for the total scale (p < 0.001).**
The Learning Styles Scale for Health Sciences Students (LS-HSS) | From enrollment to the end of treatment at 14 weeks
  was developed by Assoc. Prof. Mustafa Otrar and Elveda Kuyucak. Following expert review, the scale initially consisted of 70 items and underwent validity and reliability analyses. After item reduction procedures, 34 items were excluded due to low correlations with the intended constructs or cross-loadings on multiple factors, resulting in a final version of 36 items.
  The scale is a self-report, five-point Likert-type instrument. Due to the absence of another learning styles scale specifically developed for health sciences students, convergent validity could not be assessed. To enhance the generalizability of the findings, future studies are recommended to replicate the scale using larger and more diverse samples and to support quantitative results with qualitative research. Written permission for the use of the scale was obtained.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Konya, Konya
  - Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Konya

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Background] Koivisto JM, Haavisto E, Niemi H, Haho P, Nylund S, Multisilta J. Design principles for simulation games for learning clinical reasoning: A design-based research approach. Nurse Educ Today. 2018 Jan;60:114-120. doi: 10.1016/j.nedt.2017.10.002. Epub 2017 Oct 24. PMID 29096383
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29096383/